CLINICAL TRIAL: NCT00385775
Title: A Phase I Trial of AEG35156 Administered by 2-Hour Intravenous Infusion in Patients With Advanced Cancers
Brief Title: Study of XIAP Antisense for Advanced Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Dosing cohort (650mg) exceeded current 350mg dosing in other trials.
Sponsor: Aegera Therapeutics (Industry)
Responsible Party: Jacques Jolivet, MD, Senior VP Clinical, Aegera Therapeutics Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AEG35156-104
Record Dates: First submitted 2006-10-06; First posted 2006-10-11 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2008-08

CONDITIONS: Advanced Cancer
Keywords: Cancer; solid tumours; refractory; antisense; oligonucleotide
MeSH Terms: conditions — Neoplasms | interventions — AEG 35156

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AEG35156 — weekly IV solution infused over 2 hrs

SUMMARY:
This study is designed to find the maximum tolerated dose, safety and toxicity profile, and to identify any dose limiting toxicities of AEG35156 administered in 2-hour infusions to patients with advanced cancers.

DETAILED DESCRIPTION:
This is a Phase I study, single-arm, open-label, dose escalation study to establish the recommended dose and activity of AEG35156 administered as a 2-hour daily infusion over 3 days initially followed by weekly 2-hour intravenous infusions in patients with advanced cancers. Subjects eligible for study entry must have proven advanced or metastatic cancer refactory to conventional treatment or for which no conventional therapy exists. The starting dose will be a fixed dose of 60 mg/day with escalation by steps of 50 to 100% in successive cohorts. Approximately of 30 patients will be entered in the study to determine the maximum tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven diagnosis of advanced or metastatic cancer (including solid tumours and lymphoma)
* refractory to conventional treatment, or for which no conventional therapy exists with life expectancy of at least 12 weeks
* ECOG performance status of 0 or 1
* hematological and biochemical indices as specified within one week prior to treatment

Exclusion Criteria:

* known bleeding diathesis or concurrent treatment with anticoagulants
* primary brain tumours or brain metastases
* radiotherapy (except palliative), endocrine therapy, immunotherapy or chemotherapy during the previous four weeks (six weeks for nitrosoureas and mitomycin-C)
* all toxic manifestations of previous treatment must have resolved (excepting alopecia or certain Grade 1 toxicities)
* pregnant or lactating women
* major thoracic and/or abdominal surgery in the preceding 4 weeks
* high medical risks from non-malignant systemic disease including uncontrolled infection
* hepatitis B, C or Human Immunodeficiency Virus
* allergic history to antisense agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-06; Primary Completion 2008-10 (Estimated); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
Dose level at which AEG35156 is well tolerated based upon development of toxicities during the first cycle of therapy unless delayed or cumulative toxicity is encountered. Assessments done weekly. | 1 year

SECONDARY OUTCOMES:
Determine the impact of AEG35156 on inhibition and apoptosis in tumour biopsies or circulating tumour cells. | 1 year
Determine the occurence of XIAP knockdown in peripheral blood mononuclear cells. | 1 year
Determine the plasma pharmacokinetic profile of AEG35156. | 1 year
Determine the possible anti-tumour activity of XIAP. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Jolivet, MD, Study Director — Aegera Therapeutics Inc.
Locations (1):
- Christie Hospital NHS Trust, Manchester, United Kingdom